CLINICAL TRIAL: NCT06546059
Title: Gasdermin D Expression in Generalized Vitiligo Patients After Narrow-band Ultraviolet B Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Soheir Abdelhamid, Soheir Abdel-Hamid, principle investigator, South Valley University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVU-MED-,4-24,7,871
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Vitiligo, Generalized
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one group (Other)
  Interventions: Device: narrow band ultraviolet-B

INTERVENTIONS:
Device: narrow band ultraviolet-B — vitiligo patients will recevie twice sessions per week

SUMMARY:
The aim of this study is to:

1. Evaluate the role of tissue Gasdermin D expression using immunehistochemstry techniques in patients with generalized vitiligo and compare it with healthy controls.
2. Evaluation expression of tissue Gasdermin D using immunehistochemstry techniques in patients with generalized vitiligo after narrow band ultraviolet B therapy.
3. Determine whether there is a relationship between Gasdermin D levels and disease duration and involved body surface area (VISA) in vitiligo patients.

DETAILED DESCRIPTION:
The aim of this study is to:

1. Evaluate the role of tissue Gasdermin D expression using immunehistochemstry techniques in patients with generalized vitiligo and compare it with healthy controls.
2. Evaluation expression of tissue Gasdermin D using immunehistochemstry techniques in patients with generalized vitiligo after narrow band ultraviolet B therapy.
3. Determine whether there is a relationship between Gasdermin D levels and disease duration and involved body surface area (VISA) in vitiligo patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable vitiligo of 6 months duration,
* Both sex and ages(10-75)

Exclusion Criteria:

* pregnancy,
* lactation,
* patients under or previous phototherapy,
* patients on other immunosuppressives,
* patients receiving topical or systemic therapy like antioxidants and vitamins were kept off treatment for 2 weeks prior to recruitment into the study.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the role of tissue Gasdermin D expression using immunehistochemstry techniques in patients with generalized vitiligo and compare it with healthy controls. | three months
  1- Evaluate the role of tissue Gasdermin D expression using immunehistochemstry techniques in patients with generalized vitiligo and compare it with healthy controls.techniques in patients with generalized vitiligo and compare it with healthy controls.

SECONDARY OUTCOMES:
2- Evaluation expression of tissue Gasdermin D using immunehistochemstry techniques in patients with generalized vitiligo after narrow band ultraviolet B therapy. | three months
  2- Evaluation expression of tissue Gasdermin D using immunehistochemstry techniques in patients with generalized vitiligo after narrow band ultraviolet B therapy.
3- Determine whether there is a correlation between tissue immunehistochemstry Gasdermin D levels and disease duration and involved body surface area (VISA) in vitiligo patients. | three months
  3- Determine whether there is a correlation between tissue immunehistochemstry D levels and disease duration and involved body surface area (VISA) in vitiligo patients.